CLINICAL TRIAL: NCT02871531
Title: A Randomized Controlled Trial Comparing Pneumatic Retinopexy Versus Vitrectomy for the Management of Primary Retinal Detachment in Patients With Extended Criteria; Anatomical Success, Functional Success and Impact on Patient Quality of Life
Brief Title: Pneumatic Retinopexy Versus Vitrectomy for Retinal Detachment in Patients With Extended Criteria
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Extended criteria pneumaticPPV
Record Dates: First submitted 2016-08-11; First posted 2016-08-18 (Estimated); Last update posted 2019-08-26 (Actual); Status verified 2019-08

CONDITIONS: Rhegmatogenous Retinal Detachment
Keywords: retinal detachment; pneumatic retinopexy; vitrectomy
MeSH Terms: conditions — Retinal Detachment | interventions — Lasers; Cryotherapy; Vitrectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pneumatic retinopexy (Experimental): Patients with retinal detachment allocated to pneumatic retinopexy
  Interventions: Procedure: Pneumatic retinopexy
- Vitrectomy (Experimental): Patients with retinal detachment allocated to vitrectomy
  Interventions: Procedure: Vitrectomy

INTERVENTIONS:
Procedure: Pneumatic retinopexy
  Other Names: Pneumatic retinopexy plus laser/cryotherapy
  Arms: Pneumatic retinopexy
Procedure: Vitrectomy
  Other Names: Pars plana vitrectomy plus laser/cryotherapy
  Arms: Vitrectomy

SUMMARY:
Objective: To compare outcomes of retinal detachment repair following pneumatic retinopexy (PnR) versus pars plana vitrectomy in terms of anatomical success, functional success and patient quality of life in patients with extended criteria.

Methods: A prospective, randomized, controlled trial will be conducted with 178 patients presenting at St. Michael's Hospital with primary retinal detachment (RD). Inclusion criteria include: a single or multiple retinal tears in detached retina between 7 and 5 o'clock being of any size and any distance apart from each other, including giant retinal tears with inferior aspect above 5 and 7 o'clock, RD with no identifiable tear but where suspected tear is between 7 and 5 o'clock, retinoschisis with RD if tears are located between 7 and 5 o'clock, mild proliferative vitreoretinopathy, none or mild vitreous hemorrhage. Patients will be excluded if there is a small retinal tear or multiple tears less than 30o apart between 8 and 4 o'clock in detached retina, retinal tear in detached retina between 5 and 7 o'clock, <18 years old, inability to read English, mental incapacity, previous history of RD, scleral buckle or vitrectomy in index eye, inability to maintain appropriate head posture at post-operative period and inability to visualize peripheral retinal due to media opacity. Patients will be randomly allocated into two groups: PnR + cryotherapy/laser or vitrectomy + cryotherapy/laser and the intervention will take place within 24 hours and 72 hours for attached and detached macula status, respectively. Patients will undergo a complete ophthalmological examination, including visual acuity and fundus assessment at baseline and at 3, 6 and 12 months after surgery. Visual acuity will also be measured at 1, 7 and 30 days after surgery. Global health related quality of life will be evaluated with the SF-36v2 questionnaire at baseline, 1 month, 1 and 2 years after intervention, while the VFG25 questionnaire will be applied at 3, 6, 12 and 24 months after surgery to measure vision related quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Single retinal tear or group of tears (any distance apart) in detached retina located between 7 and 5 o'clock.
* Retinal detachment with no identifiable tear but where suspected tear is located between 7-5 o'clock based on Lincoff rules
* Any size of retinal tear, including giant retinal tears, if the inferior aspect of it is above 5 and 7 o'clock
* Retinoschisis with retinal detachment if tears are located between 7 and 5 o'clock
* There may be mild proliferative vitreoretinopathy (unless there is a visible traction on the break)
* None or mild vitreous hemorrhage. Note: vitreous hemorrhage will be considered mild if it does not impair an adequate examination of the retinal periphery.
* In the opinion of the investigator, PnR is likely to achieve anatomical re-attachment of the retina

Exclusion Criteria:

* Group of tears <30o apart in detached retina if all located within 8-4 o'clock
* Single retinal tear smaller than 1 o'clock in detached retina between 8-4 o'clock
* Retinal tears below the 5 and 7 o'clock meridian in detached retina (note that additional tears in attached retina are acceptable)
* Inability to read English language
* Age <18 years
* Mental incapacity
* Previous vitrectomy or scleral buckle (index eye)
* Previous retinal detachment (index eye)
* Inability to maintain the strict post-operative posturing requirements of pneumatic retinopexy
* Inability to carry out detailed examination of the peripheral retina due to media opacity NOTE: Lens/posterior hyaloid status does not affect eligibility.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Estimated)
Dates: Start 2016-11; Primary Completion 2021-11 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Visual acuity (ETDRS) | 12 months post intervention

SECONDARY OUTCOMES:
Visual acuity (ETDRS) | 3, 6 and 24 months post intervention
Visual acuity (Snellen) | 1 week, 1, 3, 6, 12 and 24 months post intervention
Subjective visual function (VFQ25) | 3, 6, 12 and 24 months post intervention
Anatomical success (complete retinal re-attachment with no adjuvant surgical procedure) | 3, 6, 12 and 24 months post intervention
Subjective health related quality of life (SF-36v2) | baseline, 1 month, 12 and 24 months post intervention
Aniseikonia rates | 12 and 24 months
Metamorphopsia rates | 3, 12 and 24 months
Retinal displacement rate measured with fundus autofluorescence | 3 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Rajeev Muni, FRSCS, Principal Investigator — staff; Verena Juncal, MD, Principal Investigator — research fellow
Locations (2):
- Canada (2):
  - St. Michael's Hospital Eye Clinic, Toronto, Ontario
  - Sunnybrook Health Sciences Centre, Toronto